CLINICAL TRIAL: NCT03525366
Title: Prospective Evaluation Of Outcomes For Patients Undergoing Radiofrequency Ablation (RFA) Using HALO Ultra Device For Gastric Antral Vascular Ectasia (GAVE)
Acronym: GAVE
Status: Withdrawn | Type: Observational
Why Stopped: lack of funding
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Nirav C Thosani, Assistant Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-15-0449
Record Dates: First submitted 2016-01-04; First posted 2018-05-15 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Gastric Antral Vascular Ectasia
MeSH Terms: conditions — Gastric Antral Vascular Ectasia | interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Radiofrequency ablation — Radiofrequency Ablation (RFA) as an intervention is part of standard of care at Memorial Herman Hospital, Houston.

SUMMARY:
The purpose: To determine the safety and efficacy of Radiofrequency Ablation (RFA) HALO Ultra system in patients with Gastric Antral Vascular Ectasia patient cohort (GAVE).

Research design: This is a prospective observational study. Procedure Used: Radiofrequency Ablation

Risks and potential benefits:

There are no risks associated with this study as it is a retrospective chart review. Potential benefits include the knowledge gained from this study which may be of help to patients in the future.

Importance of knowledge that may reasonably be expected to result The knowledge gained from this study may be of help to other patients in the future.

DETAILED DESCRIPTION:
The purpose of this study is to see how well study device works at treating people with Gastric Antral Vascular Ectasia (GAVE). The device has already been approved by the Food and Drug Administration (FDA) and is a part of standard of care. You have been invited to join this research study because you require diagnostic or therapeutic evaluation of the Gastric Antral Vascular Ectasia by RFA.

This is a single -site study being performed at the University of Texas Health Science Center. The study will enroll a total 1000 patients with GAVE. This study is purely observational and will collect clinical information regarding your GAVE

ELIGIBILITY:
Inclusion Criteria:

* In-patients
* Patients diagnosed with GAVE
* Patients undergoing radiofrequency ablation with HALO ULTRA device

Exclusion Criteria:

* Patients who were not diagnosed with GAVE
* Patients undergoing RFA with HALO ULTRA device for diseases other than GAVE.
* Patients with GAVE receiving other endoscopic therapies like argon plasma coagulation (APC) or radiofrequency ablation (RFA) with devices other than HALO ULTRA

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with Gastric Antral Valve Ectasia cohort undergoing radiofrequency ablation therapy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2022-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of RFA therapy sessions with the HALO ULTRA device | Up to 1 year after first RFA session with the HALO ULTRA device
  Patients will be followed up until the time that they achieve resolution of Gastric Antral Vascular Ectasia (GAVE) lesions, which may be up to 1 year.
Hemoglobin level | Before the first RFA session with HALO ULTRA device.
Hemoglobin level | At the time of resolution of GAVE lesions, which is up to 1 year after first RFA session with HALO ULTRA device.
  Hemoglobin level will be assessed at the time the patient achieves resolution of Gastric Antral Vascular Ectasia (GAVE) lesions, which may be up to 1 year.
Number of patients who require blood transfusion | Before the first RFA session with HALO ULTRA device
Number of patients who require blood transfusion | At the time of resolution of GAVE lesions, which is up to 1 year after first RFA session with HALO ULTRA device.
  Patients will be followed up until the time that they achieve resolution of Gastric Antral Vascular Ectasia (GAVE) lesions, which may be up to 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Nirav Thosani, MD MHA, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States